CLINICAL TRIAL: NCT01543620
Title: Prospective Observational Study to Evaluate Biomarkers of Aminoglycoside Nephrotoxicity in Patients With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Foundation for the National Institutes of Health (Other)
Collaborators: University of Southern California (Other); University of Minnesota (Other); M.D. Anderson Cancer Center (Other); Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Amgen (Industry); AstraZeneca (Industry); Eli Lilly and Company (Industry); Johnson & Johnson (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); Critical Path Institute (Unknown); Predictive Safety Testing Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: Kidney Safety - Aminoglycoside
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-07

CONDITIONS: Cystic Fibrosis
Keywords: kidney safety; biomarkers; serum creatinine; BUN; cystic fibrosis; head and neck cancer; renal injury; drug induced acute kidney injury; aminoglycoside; cisplatin; nephrotoxicity; biomarker qualification
MeSH Terms: conditions — Cystic Fibrosis; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with cystic fibrosis treated with aminoglycosides
- Patients with cystic fibrosis not treated with aminoglycosides

SUMMARY:
The project is designed to test new biomarkers that are more sensitive than the current standard in detecting injury to the proximal kidney tubule and will establish better criteria for when kidney safety concerns may halt further testing of a drug in humans.

DETAILED DESCRIPTION:
The goal of this clinical study is to advance the acceptance of new biomarkers designed to detect drug-induced kidney injury in clinical trials.

The Kidney Safety Project is being conducted at four major medical centers:

* University of Southern California
* University of Minnesota
* MD Anderson Cancer Center
* Dana-Farber Cancer Institute.

Blood and urine samples will be collected from patients undergoing treatment with either cisplatin or aminoglycosides, which are two different drugs known to cause injuries to the proximal tubule of the kidney. Aminoglycosides are a common antibiotic drug taken by patients with cystic fibrosis. Cisplatin is a common chemotherapy drug taken by patients with head and neck cancer.

The Aminoglycoside Study of the Kidney Safety Project is being conducted at the University of Southern California and the University of Minnesota and aims to evaluate aminoglycoside induced acute kidney injury in patients with cystic fibrosis.

The companion study, the Cisplatin Study of the Kidney Safety Project, is being conducted at the MD Anderson Cancer Center and the Dana-Farber Cancer Institute and aims to evaluate cisplatin induced acute kidney injury in patients with head and neck cancer.

The data from the Kidney Safety Project, from both the Aminoglycoside Study and the Cisplatin Study, will be combined for determination of the best biomarkers for predicting drug-induced acute kidney injury.

ELIGIBILITY:
Inclusion criteria:

1. Males and females ≥ 18 years of age.
2. Documentation of CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   * Sweat chloride greater than or equal to 60 mEq/L by quantitative pilocarpine iontophoresis test.
   * Two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene; or
   * Abnormal nasal potential difference.
3. Hospitalized and initiated on systemic antibiotic therapy for treatment of an acute pulmonary exacerbation.
4. Willingness and ability to comply with study procedures and study restrictions.
5. Ability to provide written informed consent.

Exclusion criteria:

1. Chronic kidney disease defined by microalbuminuria (> 30 mcg/mg creatinine) or eGFR < 60 mL/min/1.73m2.
2. Receiving medications known to alter the tubular secretion of creatinine (e.g. trimethoprim, cimetidine).
3. Hospitalized for treatment of an acute pulmonary exacerbation or received intravenous aminoglycoside antibiotics within 3-months of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cystic fibrosis patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beringer, PharmD, Principal Investigator — University of Southern California; Joanne Billings, MD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - University of Minnesota - Cystic Fibrosis Center, Minneapolis, Minnesota
  - University of Utah, Salt Lake City, Utah